CLINICAL TRIAL: NCT06721403
Title: Assessment of Anxiety,Depressive Symptoms &PTSD in Cases of Post Ectopic Pregnancy
Brief Title: Psychatric Effect of Ectopic Pregnancy
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marina Reda Youssef, Assistant lecture, Assiut University
Other Study IDs: Anxiety post ectopic pregnancy
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Ectopic Pregnancy
MeSH Terms: conditions — Pregnancy, Ectopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
Assessment of anxiety,depressive symptoms and post traumatic stress after ectopic pregnancy Determine factors associated with development of anxiety,depressive symptoms and post-traumatic stress after ectopic pregnancy

DETAILED DESCRIPTION:
Ectopic pregnancy is any pregnancy in which the fertilized ovum implants outside the intrauterine cavity. More than 95 percent of ectopic pregnancies occur in the fallopian tubes.

Another 2.5 percent occur in the cornua of the uterus, and the remainder are found in the ovary, cervix or abdominal cavity.

Ectopic pregnancy causes major maternal morbidity and mortality, with pregnancy loss, and its incidence is increasing worldwide.

Previous ectopic pregnancy becomes a more significant risk factor with each successive occurrence. With one previous ectopic pregnancy treated by linear salpingostomy, the recurrence rate ranges from 15 to 20 percent, depending on the integrity of the contralateral tube.

The unanticipated and sudden loss of a pregnancy can be a devastating and traumatic experience resulting in high levels of psychological morbidity for some women.

EPLs can significantly contribute to the overall burden of psychopathology within a population. Recognition of this impact is important, so that severely affected individuals may be screened and treated appropriately. Further research to establish risk factors to promptly identify and treat these patients, and to optimize their management, is crucial"

ELIGIBILITY:
Inclusion Criteria:

* All pregnant woman 18:45 years old presented with ectopic pregnancy.

Exclusion Criteria:

* intrauterine pregnancy
* previous diagnosis of psychiatric disorders
* Unwell to give consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All pregnant women 18:45 years old presented with ectopic pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Effect of ectopic pregnancy | Within one week
  Prevalence of anxiety,depressive symptoms and post-traumatic stress disorder after ectopic pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abbas, Prof, Study Director — Assiut University

REFERENCES:
- [Background] Farren J, Jalmbrant M, Ameye L, Joash K, Mitchell-Jones N, Tapp S, Timmerman D, Bourne T. Post-traumatic stress, anxiety and depression following miscarriage or ectopic pregnancy: a prospective cohort study. BMJ Open. 2016 Nov 2;6(11):e011864. doi: 10.1136/bmjopen-2016-011864. PMID 27807081